CLINICAL TRIAL: NCT06975033
Title: The Impact of Discharge Educational Discharge Videos on Post-Operative Care Utilization After Holmium Laser Enucleation of the Prostate (HoLEP) Procedures
Brief Title: The Impact of an Educational Discharge Video on Post-Operative Health Care Utilization After Holmium Laser Enucleation of the Prostate (HoLEP) Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: State University of New York - Upstate Medical University (Other); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-43311
Record Dates: First submitted 2025-04-04; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: HoLEP; Patient Satisfaction; Educational Video Intervention
MeSH Terms: conditions — Patient Satisfaction | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Experimental): Participants will watch video.
  Interventions: Other: Video
- No Video (No Intervention): Participants will not watch video.

INTERVENTIONS:
Other: Video — Participants will watch video.
  Arms: Video

SUMMARY:
This will be a randomized interventional study. Patients scheduled to undergo a HoLEP at UCSF will be randomized into two groups after the procedure: one group will watch a scripted educational HoLEP video and the other group will not receive a video. We will monitor the post-operative care utilization after discharge. Secondary outcomes will include patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18+
2. Patients scheduled for a HoLEP procedure
3. Patients willing to complete both baseline and follow up surveys
4. Patients able to provide informed consent
5. Patients are English-speaking and understand English

Exclusion Criteria:

1. Patients under 18+
2. Patients unable to consent
3. Patients unable to complete surveys
4. Patients without a prostate.
5. Patients are non-English speakers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Healthcare Utilization | up to 60 days (estimated time frame between initial surgery and first follow up visit)
  Healthcare utilization will include MyChart messages, phone calls to clinic, unscheduled clinic visits, emergency/urgent care visits, etc.
Participant Satisfaction | up to 60 days (estimated time frame between initial surgery and first follow up visit)
  Patients will complete a patient satisfaction survey .This survey ranges from 1 (strongly agree) to 5 (strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: David Bayne, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - University of Rochester Medical Center, Rochester, New York
  - Scott SUNY Upstate Medical University, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No